CLINICAL TRIAL: NCT02814617
Title: The Efficacy and Safety of Cordyceps Sinensis Mycelium Culture Extract(Paecilomyces Hepiali, CBG-CS-2) on Promotion of Immunity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CBG-PI-CME
Record Dates: First submitted 2016-06-14; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Immunity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cordyceps sinensis mycelium culture extract (Experimental): Cordyceps sinensis mycelium culture extract 1.68 g
  Interventions: Dietary Supplement: Cordyceps sinensis mycelium culture extract 1.68 g
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cordyceps sinensis mycelium culture extract 1.68 g — Cordyceps sinensis mycelium culture extract 1.68 g
  Arms: Cordyceps sinensis mycelium culture extract
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The investigators performed randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Cordyceps sinensis mycelium culture extract (Paecilomyces hepiali, CBG-CS-2) on promotion of immunity. The investigators measured promotion of immunity parameters , including Cytotoxicity, Cytokine (IL-1β, IL-2, IL-4, IL-10, IL-12, IFN-γ, TNF-α).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 20-75 years old
* Able to give informed consent

Exclusion Criteria:

* WBC concentration below 3000 ㎕, over 8000㎕
* Subjects with BMI < 18.5 kg/m2 at screening visit
* Allergic or hypersensitive to any of the ingredients in the test products
* Diagnosed of gastrointestinal disease such as Immune-related diseases, severe hepatic, renal failure, and diabetes
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in serum natural killer cell activity | Baseline, 8 weeks

SECONDARY OUTCOMES:
Changes in Cytokine(IL-1β, IL-2, IL-4, IL-10, IL-12, IFN-γ, TNF-α) | Baseline, 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Jung SJ, Jung ES, Choi EK, Sin HS, Ha KC, Chae SW. Immunomodulatory effects of a mycelium extract of Cordyceps (Paecilomyces hepiali; CBG-CS-2): a randomized and double-blind clinical trial. BMC Complement Altern Med. 2019 Mar 29;19(1):77. doi: 10.1186/s12906-019-2483-y. PMID 30925876